CLINICAL TRIAL: NCT04276584
Title: Effect of Speaking Aloud vs. Positive Expiratory Pressure Therapy on Oxygen Saturation After Abdominal Surgery.
Brief Title: Effect of Speaking Aloud After Abdominal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201822831
Record Dates: First submitted 2020-02-10; First posted 2020-02-19 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Respiratory Complications
Keywords: abdominal surgery; hypoxia; lung function; ventilation; Carbon dioxide partial pressure; oxygen situation; Postoperative; Positive expiratory pressure therapy
MeSH Terms: conditions — Hypoxia; Respiratory Aspiration | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Positive expiratory pressure is given to patients after abdominal surgery in order to improve postoperative oxygen saturation and lung function. We aim to test whether speaking loudly from a given text improve postoperative oxygen saturation and ventilation. 50 patients will be investigated in a randomized controlled trial with cross-over design starting either with positive expiratory pressure therapy (10 times 3 inspiration and expiration to positive expiratory pressure) or with speaking loudly from a given text.
Who Masked: Outcomes Assessor
Masking Description: Patients are given a serial number. The randomization orders are blinded to the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive expiratory pressure (Active Comparator): Deep inspiration followed by expiration to a resistance of 10-15 cm of water pressure. Done three times, each time with 10 inspiration/expiration cycles
  Interventions: Device: Positive expiratory pressure
- Speaking loudly (Experimental): Speaking loudly during 3 minutes.
  Interventions: Other: Speaking loudly during about 3 minutes

INTERVENTIONS:
Device: Positive expiratory pressure — Three blocks of 10 deep inspiration followed by expiration against a positive airway pressure device of 10-15 cm of water pressure. Repeated three times. Estimated time of 3 minutes time.
  Arms: Positive expiratory pressure
Other: Speaking loudly during about 3 minutes — A specified swedish text
  Arms: Speaking loudly

SUMMARY:
Hypoxia and reduced vital capacity is commonly occurring after abdominal surgery. Positive expiratory pressure is one treatment suggested to improve lung function after surgery. We aim to test whether speaking improves postoperative oxygen saturation and ventilation after abdominal surgery. In a cross-over design, 50 subjects will be randomized to start with either positive expiratory pressure maneuvers, i.e. deep inspiration followed by expiration in a positive expiratory pressure device at 10-15 cm of water, or to start with reading a text loudly. Arterial blood gases will be taken at study start. Patients will be monitored using Noxturnal T3, Res Med for respiration and pulse oximetry, and online transcutaneous carbon dioxide partial pressure measurements (SenTec Digital monitoring systems). Main outcome measurements include oxygen saturation after speaking compared with positive expiratory pressure therapy.

DETAILED DESCRIPTION:
Hypoxia and reduced vital capacity is commonly occurring after abdominal surgery. Positive expiratory pressure is one treatment suggested to improve lung function after surgery, but there is a lack of evidence of effect. En passant, we observed that oxygen saturation was improved when patients talked postoperative day 1. We aim to test whether speaking improves postoperative oxygen saturation and ventilation after abdominal surgery.

It was estimated that a sample size of 34 patients was needed to detect a mean and (SD) difference in oxygen saturation of 1% (2%) and to detect a difference in transcutaneous carbon dioxide partial pressure of 0.5 kPa (1 kPa) with a significance level of 0.05 and a power of 0.8.

In a randomized controlled trial, 50 subjects will be randomized (1:1) to start with either positive expiratory pressure maneuvers, i.e. 3 x 10 deep inspiration followed by expiration in a positive expiratory pressure device of 10-15 cm H20 or to start with reading a text loudly during 3 minutes. Patients will be monitored using Noxturnal T3, Res Med for respiration and pulse oximetry. SenTec Digital Monitoring systems for online transcutaneous carbon dioxide partial pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Performed abdominal surgery within 2 days at the departments of surgery, urology or gynecology at Umeå university hospital

Exclusion Criteria:

* Patients referred to ICU because of immediate postoperative complications.

  * Patients who are unable to perform the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation after speaking aloud | At day 1 or 2 after surgery
  Oxygen saturation (SaO2) at 7 minutes after speaking aloud compared with positive expiratory pressure therapy

SECONDARY OUTCOMES:
Ventilation after speaking aloud | At day 1 or 2 after surgery
  Transcutaneous carbon dioxide partial pressure after speaking aloud compared with positive expiratory pressure therapy

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, Prof, Principal Investigator — Dept Surgical and periopertive sciences, Umeå university, Sweden
Locations (1):
- Dept of Surgery, Inst of Surgical and Perioperative sciences, Umeå, Umea, Sweden

IPD SHARING:
Plan to Share IPD: Yes
To share all the measured data from each participant.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the study is published and 10 years forward
Access Criteria: Deidentified individual participant data will be available to medical researchers by request in accordance with local registration and ethical approval when the article has been published until December 2031. All proposals requesting data access will be reviewed on a case by case basis and will need to specify an analysis plan and will need approval of the scientific board before any data can be released.